CLINICAL TRIAL: NCT01961336
Title: The Effect of Transdermal Testosterone Pretreatment in Poor Responders Undergoing Ovarian Stimulation for In-vitro Fertilization (IVF)
Brief Title: Transdermal Testosterone Pretreatment in Poor Responders Undergoing IVF
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Aristotle University Of Thessaloniki (Other)
Collaborators: University of Thessaly (Other)
Responsible Party: Principal Investigator, E.M. Kolibianakis, Assistant Professor, Aristotle University Of Thessaloniki
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UHR-9
Record Dates: First submitted 2013-10-10; First posted 2013-10-11 (Estimated); Last update posted 2016-06-28 (Estimated); Status verified 2016-06

CONDITIONS: Subfertility
Keywords: IVF, poor responder, testosterone
MeSH Terms: conditions — Infertility | interventions — Testosterone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Testosterone (Experimental): Long depot follicular GnRH agonist protocol. On day 21 initiation of ovarian stimulation with recombinant FSH for ICSI. If necessary downregulation will be achieved with additional daily agonist s.c.
  10 mg of testosterone gel applied on the external side of the thigh for 21 days starting from the first day of menstruation prior to initiation of ovarian stimulation with rFSH for IVF/ICSI.
  Interventions: Drug: Testosterone
- Control (No Intervention): Long depot follicular GnRH agonist protocol. On day 21 initiation of ovarian stimulation with recombinant FSH for ICSI. If necessary downregulation will be achieved with additional daily agonist s.c.

INTERVENTIONS:
Drug: Testosterone — 10 mg of testosterone gel applied on the external side of the thigh for 21 days starting from the first day of menstruation prior to initiation of ovarian stimulation with rFSH for IVF/ICSI
  Arms: Testosterone

SUMMARY:
Ιt has been suggested that the accumulation of androgens in the micro milieu of the primate ovary, plays a critical role in early follicular development and granulosa cell proliferation. Increased intraovarian concentration of androgens seems to augment follicle stimulating hormone (FSH) receptor expression in granulosa cells and thus, potentially leading to enhanced responsiveness of ovaries to FSH. In addition, androgen excess has been shown to stimulate early stages of follicular growth and increase the number of pre-antral and antral follicles.

On the basis of these data, it has been hypothesized that increasing androgen concentration in the ovarian micro milieu in poorly responding patients might lead to an increase in the number and the maturity of oocytes after ovarian stimulation for IVF. Hence, recent efforts have been focused on the potential benefit of androgen administration in the probability of pregnancy in poor responders undergoing ovarian stimulation for IVF.

Pretreatment with transdermal testosterone has been suggested as a safe and effective way of increasing the intraovarian androgen concentration. Recently, published, randomized control trials (RCTs) have evaluated transdermal testosterone in poor responders undergoing ovarian stimulation for IVF, with inconclusive results.

In view of the conflicting or inconclusive data regarding the efficacy of the proposed intervention, this study will attempt to explore the role of transdermal testosterone pretreatment in poor responders undergoing IVF through a properly designed RCT. The lack of a universal definition of poor responders has been identified previously and recently, in an attempt to address this issue, universal criteria for the definition of poor ovarian response have been proposed following a consensus meeting in Bologna. In the present study, the Bologna criteria will be used on the contrary to previous studies.

Despite the advancement in assisted reproduction technologies, poor ovarian response (POR) is still considered to be one of the most challenging tasks in reproductive medicine. Poor ovarian response is considered to be an inadequate response to ovarian stimulation, defined usually by a low number of oocytes retrieved or a low number of developing follicles in a previous or in the running, respectively, in vitro fertilization (IVF) cycle. Given the severely diminished probability of pregnancy after IVF in these patients, the identification of an indisputably efficacious treatment, such as testosterone pretreatment, would be a promising alternative for poor responders undergoing IVF.

ELIGIBILITY:
Inclusion Criteria:

* Advanced maternal age (≥40 years) or any other risk factor for POR
* A previous POR (≤3 oocytes with a conventional stimulation protocol)
* An abnormal ovarian reserve test (i.e. AFC < 5-7 follicles or AMH < 0.5- 1.1 ng/ml)

Exclusion Criteria:

* History of previous ovarian surgery
* Women with endocrine or metabolic disorders
* Women with active cancer disease
* Women with Stage III-IV Endometriosis
* Women with known hypersensitivity or allergy in any of the components of the drug
* Sperm only by ejaculation and not from FNA, TESE or refrigeration

Min Age: 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-10; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Total number of retrieved oocytes | 36 h after triggering of final oocyte maturation

SECONDARY OUTCOMES:
Clinical pregnancy rate (evidence of intrauterine sac with fetal heart activity at 6-8 weeks of gestation) | At 6-8 weeks of gestation
Proportion of patients reaching embryo transfer | 2 days following oocyte retrieval

CONTACTS AND LOCATIONS:
Overall Officials: Efstratios M Kolibianakis, MD, MSc, PhD, Principal Investigator — Unit for Human Reproduction, 1st Dept. of Obstetrics and Gynaecology, Medical School, Aristotle University of Thessaloniki
Locations (1):
- Unit for Human Reproduction, 1st Dept of Obstetrics and Gynaecology, Medical School, Aristotle University of Thessaloniki, Thessaloniki, Greece

REFERENCES:
- [Derived] Bosdou JK, Venetis CA, Dafopoulos K, Zepiridis L, Chatzimeletiou K, Anifandis G, Mitsoli A, Makedos A, Messinis IE, Tarlatzis BC, Kolibianakis EM. Transdermal testosterone pretreatment in poor responders undergoing ICSI: a randomized clinical trial. Hum Reprod. 2016 May;31(5):977-85. doi: 10.1093/humrep/dew028. Epub 2016 Mar 7. PMID 26956551